CLINICAL TRIAL: NCT00354107
Title: A Phase I/II Pilot Study of Ifosfamide, Carboplatin and Etoposide Therapy (ICE) and SGN-30 (NSC# 731636, IND#) in Children With CD30+ Recurrent Anaplastic Large Cell Lymphoma
Brief Title: Ifosfamide, Carboplatin, Etoposide, and SGN-30 in Treating Young Patients With Recurrent Anaplastic Large Cell Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00407; NCI-2009-00407 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ANHL06P1; CDR0000486425; ANHL06P1 (Other: Children's Oncology Group); ANHL06P1 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Results first posted 2014-01-01 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-02

CONDITIONS: Anaplastic Large Cell Lymphoma; Recurrent Childhood Anaplastic Large Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic | interventions — SGN-30 monoclonal antibody; Brentuximab Vedotin; Hydrocortisone; Ifosfamide; indolepropanol phosphate; Carboplatin; Etoposide; Methotrexate; merphos; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (monoclonal antibody therapy, chemotherapy) (Experimental): Patients receive monoclonal antibody SGN-30 IV alone on day 1 in weeks 1-8. Beginning in week 5, patients receive ICE chemotherapy comprising ifosfamide IV over 2 hours on days 1-3, carboplatin IV over 1 hour on day 1, and etoposide IV over 1 hour on days 1-3. Treatment with ICE repeats every 3 weeks for 6 courses** in the absence of unacceptable toxicity. Patients also receive intrathecal therapy comprising methotrexate, cytarabine, and hydrocortisone once on day 29 (week 5).
  Cohorts of 3-6 patients receive a pre-determined dose of monoclonal antibody SGN-30 with possible dose de-escalation to 1 dose level below in the event of ≥ 2 of 6 patients experience dose-limiting toxicity (DLT). The dose at which ≤ 1 of 6 patients experience DLT will be used in a phase II study.
  Interventions: Biological: monoclonal antibody SGN-30; Drug: therapeutic hydrocortisone; Drug: ifosfamide; Drug: carboplatin; Drug: etoposide; Drug: methotrexate; Drug: cytarabine; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: monoclonal antibody SGN-30 — Given IV
  Other Names: SGN-30
Drug: therapeutic hydrocortisone — Given IT
  Other Names: Aeroseb-HC; Barseb HC; Cetacort; Cort-Dome; Cortef
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: methotrexate — Given IT
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: cytarabine — Given IT
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of SGN-30 when given together with ifosfamide, carboplatin, and etoposide and to see how well they work in treating young patients with recurrent anaplastic large cell lymphoma. Drugs used in chemotherapy, such as ifosfamide, carboplatin, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as SGN-30, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Define and describe the toxicities of monoclonal antibody SGN-30 alone (window) and in combination with ifosfamide, carboplatin, and etoposide (ICE) in pediatric patients with CD30-positive recurrent anaplastic large cell lymphoma.

II. Define, preliminarily, the antitumor activity of monoclonal antibody SGN-30 alone (window) and in combination with ICE in these patients.

SECONDARY OBJECTIVES:

I. Characterize the pharmacokinetics of monoclonal antibody SGN-30 in these patients.

II. Characterize the soluble CD30 concentrations at time of relapse in these patients.

III. Characterize the development of human antichimeric antibodies in these patients.

IV. Measure minimal residual disease in these patients.

OUTLINE: This is a multicenter, pilot, phase I, dose-finding study of monoclonal antibody SGN-30 followed by a phase II study.

Patients receive monoclonal antibody SGN-30 IV alone on day 1 in weeks 1-8. Beginning in week 5, patients receive ICE chemotherapy comprising ifosfamide IV over 2 hours on days 1-3, carboplatin IV over 1 hour on day 1, and etoposide IV over 1 hour on days 1-3. Treatment with ICE repeats every 3 weeks for 6 courses** in the absence of unacceptable toxicity. Patients also receive intrathecal therapy comprising methotrexate, cytarabine, and hydrocortisone once on day 29 (week 5).

NOTE: **Patients planning to undergo bone marrow transplantation (BMT) receive 2 courses of ICE only and then undergo BMT off study.

Cohorts of 3-6 patients receive a pre-determined dose of monoclonal antibody SGN-30 with possible dose de-escalation to 1 dose level below in the event of ≥ 2 of 6 patients experience dose-limiting toxicity (DLT). The dose at which ≤ 1 of 6 patients experience DLT will be used in a phase II study.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed anaplastic large cell lymphoma
* CD30-positive disease
* Must be in first or second relapse
* Measurable disease
* No CNS disease
* Karnofsky performance status (PS) 60-100% (> 16 years of age) OR Lansky PS 60-100% (≤ 16 years of age)
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³ (transfusion independent)

  * Platelet count ≥ 20,000/mm³ if bone marrow involvement (platelet transfusions allowed)
* Hemoglobin ≥ 8.0 g/dL (RBC transfusion independent, unless bone marrow involvement)
* Creatinine adjusted according to age as follows:

  * No greater than 0.4 mg/dL (≤ 5 months)
  * No greater than 0.5 mg/dL (6 months-11 months)
  * No greater than 0.6 mg/dL (1 year-23 months)
  * No greater than 0.8 mg/dL (2 years-5 years)
  * No greater than 1.0 mg/dL (6 years-9 years)
  * No greater than 1.2 mg/dL (10 years-12 years)
  * No greater than 1.4 mg/dL (13 years and over [female])
  * No greater than 1.5 mg/dL (13 years to 15 years [male])
  * No greater than 1.7 mg/dL (16 years and over [male])
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT < 3 times ULN
* Albumin ≥ 2 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No evidence of graft-vs-host disease
* No documented active infection requiring antibiotics
* No isolated bone recurrence
* Recovered from prior therapy
* At least 3 months since prior monoclonal antibody therapy
* At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas)
* At least 7 days since prior hematopoietic growth factor therapy
* At least 3 months since prior biologic (antineoplastic) agents
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 3 months since prior total-body irradiation, craniospinal radiotherapy, or radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow irradiation
* At least 2 months since prior stem cell transplantation or rescue
* No prior monoclonal antibody SGN-30
* Concurrent steroids allowed provided dose has been stable or decreasing for the past 7 days
* No concurrent immunosuppressive agents
* No concurrent dexamethasone as an antiemetic
* No other concurrent investigational drug or anticancer agents, including chemotherapy, radiotherapy, immunotherapy, or biological therapy

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Sandlund, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Monoclonal Antibody Therapy, Chemotherapy): Patients receive monoclonal antibody SGN-30 (dosage 12mg/kg) IV alone on day 1 in weeks 1-8. Beginning in week 5, patients receive ICE chemotherapy comprising ifosfamide IV (dosage 3g/m2) x 3 days over 2 hours on days 1-3, carboplatin IV (635mg/m2) over 1 hour on day 1, and etoposide IV (dosage 100/m2) over 1 hour on days 1-3. Treatment with ICE repeats every 3 weeks for 6 courses** in the absence of unacceptable toxicity. Patients also receive intrathecal therapy (dosage dependent on age) comprising methotrexate, cytarabine, and hydrocortisone once on day 29 (week 5).
  Cohorts of 3-6 patients receive a pre-determined dose of monoclonal antibody SGN-30 with possible dose de-escalation to 1 dose level below (dosage 8mg/kg) in the event of ≥ 2 of 6 patients experience dose-limiting toxicity (DLT). The dose at which ≤ 1 of 6 patients experience DLT will be used in a phase II study.
Period: Overall Study
Arm/Group | Treatment (Monoclonal Antibody Therapy, Chemotherapy)
Started | 5
Completed | 0
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Monoclonal Antibody Therapy, Chemotherapy)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 5655 [3157 to 5786]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4
  Jordan | 1

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Anti tumor activity as assessed by computed tomography of neck/chest/abdomen/pelvis, positron emission tomography scan and/or gallium scan. Assessed by physical examination appropriate imaging studies. Bone marrow aspirate/biopsy must be normal and any macroscopic nodules in any organs detectable on imaging techniques should no longer be present. Gallium scans must be negative if initially positive.
Time Frame: Week 4
Measure: Number; unit: percent
Arm/Group | Treatment (Monoclonal Antibody Therapy, Chemotherapy)
Number analyzed (Participants) | 4
percent | 50

2. Secondary Outcome: Pharmacokinetics of Monoclonal Antibody SGN-30 Assessed by Enzyme-linked Immunosorbent Assay (ELISA) Methods
Time Frame: At baseline, at weeks 1, 2, 5, 6, and 11
Population: These data were not collected to assess this study aim and will never be reported.
Arm/Group | Treatment (Monoclonal Antibody Therapy, Chemotherapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: CD30 Concentrations Levels as Assessed by ELISA
Description: Summarized using appropriate descriptive statistics and reported with associated exact 95% confidence intervals. Although the limited sample size precludes formal hypothesis testing, exploratory analysis of the association between soluble CD30 levels and PK parameters and response will be performed.
Time Frame: At baseline
Population: These data were not collected to assess this study aim and will never be reported.
Arm/Group | Treatment (Monoclonal Antibody Therapy, Chemotherapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Development of Human Antichimeric Antibodies by Using ELISA Method
Description: Change in level from baseline to week 11 will be summarized using appropriate descriptive statistics and reported with associated exact 95% confidence intervals.
Time Frame: Change from baseline to week 11
Population: These data were not collected to assess this study aim and will never be reported.
Arm/Group | Treatment (Monoclonal Antibody Therapy, Chemotherapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Minimal Residual Disease by Using Southern Blotting or by Real-time Polymerase Chain Reaction (PCR)
Description: NPM-ALK expression will be summarized using appropriate descriptive statistics and reported with associated exact 95% confidence intervals.
Time Frame: At baseline and weeks 5 and 11
Population: These data were not collected to assess this study aim and will never be collected.
Arm/Group | Treatment (Monoclonal Antibody Therapy, Chemotherapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Monoclonal Antibody Therapy, Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Monoclonal Antibody Therapy, Chemotherapy) (N=5)
Ascites (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Monoclonal Antibody Therapy, Chemotherapy) (N=5)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Number of participants analyzed = 4. One patient was not evaluable for response. The Secondary Outcome measures will never be reported as data were not collected to assess these study aims.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less